CLINICAL TRIAL: NCT03541226
Title: Clinical Monitoring, MRI and Neuro-Ophthalmology of a Cohort of Patients With a Clinically Isolated Syndrome
Brief Title: Clinical Monitoring, MRI and Neuro-Ophthalmology of a Cohort of Patients With a Clinically Isolated Syndrome (CIS)
Acronym: cinocis
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2012_56; 2013-A00475-40 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2018-05-17; First posted 2018-05-30 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Clinically Isolated Syndrome; Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to develop tools to detect, measure, monitor and predict axonal damage in the course of CIS and during Multiple sclerosis (MS), in order to be able to consider as early as possible an adaptation of the background treatment in patients with MS. patients with radiological criteria of poor long-term clinical course.

ELIGIBILITY:
Inclusion Criteria:

* Any patient who has had a CIS of less than 4 months (+/- 15 days), with at least 1 inflammatory lesion on his initial brain MRI or with normal brain MRI associated with the presence of oligoclonal bands in the CSF,

Exclusion Criteria:

* Atypical CIS for a first relapse of multiple sclerosis (extensive myelitis, bilateral retrobulbar optic neuritis immediately)
* CIS dating more than 4 months (+/- 15 days)
* Corticotherapy in the last 4 weeks

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: patient with clinically isolated syndrome (CIS)
Sampling Method: Non-Probability Sample
Enrollment: 134 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2024-01 (Actual); Study Completion 2024-01 (Actual)

PRIMARY OUTCOMES:
severity of the disease defined by Expanded Disability Status Scale (EDSS) ≥ 2.0 | At 5 years

SECONDARY OUTCOMES:
Occurrence of a second push | At 5 years
Occurrence of progression of the EDSS (Expanded Disability Status Scale) score | At 5 years
  The scale evaluated the pyramidal, cerebellar, sensory, visual and mental functions . These make it possible to obtain a quotation between 0 and 10. The walk is called "normal" from 0 to 3.5. The walk is hampered from 4 and impossible from 7.5. The coast of 10 corresponds to the death of the patient.
  This measure differentiates two groups: severe EDSS and non-severe EDSS group,
Occurrence of a handicap objectified by the Multiple Sclerosis Functional Composite(MSFC) | At 5 years
variation of parameters measuring axonal pain / degeneration in MRI | At 5 years
variation of parameters measuring axonal pain / degeneration in OCT | At 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Outteryck, MD, PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Roger Salengro, CHRU de Lille, Lille, France

IPD SHARING:
Plan to Share IPD: No